CLINICAL TRIAL: NCT04473638
Title: Deltoid Ligament Arthroscopic Repair in Ankle Fractures: Case Series
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Nacime Salomão Barbachan Mansur, Principal Investigator, Federal University of São Paulo
Other Study IDs: Arthroscopic_Deltoid_Fx_EPM
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Ankle Injuries; Ankle Fractures; Deltoid Ligament; Sprain (Strain) (Ankle); Ligament Rupture
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic: Deltoid Arthroscopic Repair in Ankle Fractures
  Interventions: Procedure: Arthroscopic Deltoid Repair

INTERVENTIONS:
Procedure: Arthroscopic Deltoid Repair — . A 4.5 mm arthroscopic set was used to clean the joint and assess medial and associated injuries. After deltoid injury confirmation through the method already mentioned, the medial gutter was prepared. The ideal positioning for the bone anchor in the medial malleolus followed Vega's recommendations and was located in the inferolateral quadrant created by the intersection of two lines: (1) tibia-talar joint line and (2) tangent line to the medial malleolus joint surface.(14). Sutures were passed respecting the safe zone illustrated by Acevedo at al, at the area between the posterior tibial tendon and the saphenous vein (16-25mm) (15). Sutures were passed but not tightened.

SUMMARY:
To demonstrate the functional results of patients with ankle fractures operated with arthroscopic deltoid repair.

DETAILED DESCRIPTION:
Introduction: The diagnosis and treatment of ankle medial ligament lesions in malleolar fractures have always been surrounded by controversies. Even in the certainty of deltoid involvement and its consequent instability, the direct repair of this structure is not a consensus. In recent years, the arthroscopic technique to approach this ligament has been described with the objective of potentiating clinical results and minimizing possible complications.

Objective: To demonstrate the functional results of patients with ankle fractures operated with arthroscopic deltoid repair.

Methods: This is a retrospective study in patients diagnosed with ankle fractures associated with acute deltoid injuries and submitted to a malleolar fixation and deltoid arthroscopic repair between January 2018 and January 2020. All patients will fill an epidemiological questionnaire and will be evaluated for pain and function according to the Visual Analogue Scale (VAS) and the American Orthopaedic Foot and Ankle Society Score (AOFAS) at 12 months (6-24 months) average of follow-up.

Discussion: The inclusion of the deltoid complex and the low invasiveness of this technique can improve the clinical outcomes of these patients. Additional studies, with a prospective and comparative methodology are required to sustain this proposal.

ELIGIBILITY:
Inclusion Criteria:

- acute (less than two weeks) ankle fracture containing a medial ligament injury suspicion will be included. Syndesmotic lesion with a deltoid association will also be addressed

Exclusion Criteria:

* previous surgery
* autoimmune diseases
* neuropathy
* inflammatory diseases
* radiographic preoperative findings of ankle arthritis
* open medial wound
* coagulopathies
* any other condition that would contraindicate surgery

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary/Quaternary hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society - Hindfoot Score (AOFAS) | Time Frame: 6th post-operative month
  Functional Score (0 to 100 | 100 best score possible | 0 worst score possible)

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Time Frame: 6th post-operative month
  Pain Score (0 to 10 | 10 worst score possible | 0 best score possible)
Number of Complications related to Treatment | 6th post-operative month
  Complications were established as dehiscence, neural damage, infection, and re-rupture. Dehiscence was set inability to heal the soft tissue coverage until the end of the 4th post-operative week. Peripherical nerve damage defined as hypoesthesia or paresthesia not solved until the end of the 6th month after the surgery. Infection termed as clinical signs infection or pus drainage at the wound that required the use of antibiotics. Re-rupture classified as an ankle sprain event during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Nacime Salomão Barbachan Mansur, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
According to the ICMJE data sharing police, core records will be shared at an online depository and available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After article publication.
Access Criteria: A formal requisition will be needed, directly addressed to the main researcher. A good scientific reason must be included.